CLINICAL TRIAL: NCT01632514
Title: Correction of Vitamin D Deficiency to Prevent Postoperative Hypocalcemia After Thyroidectomy
Brief Title: Vitamin D Deficiency and Postoperative Hypocalcemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Debora Lucia Seguro Danilovic, M.D., PhD., University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USaoPauloGH 8624
Record Dates: First submitted 2012-06-26; First posted 2012-07-03 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Hypocalcemia
Keywords: hypocalcemia; vitamin D deficiency; cholecalciferol; thyroidectomy
MeSH Terms: conditions — Hypocalcemia; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vitamin D deficiency treatment (Active Comparator): subjects with 25OHD < 20 ng/mL that will receive 100,000U of cholecalciferol weekly for 4 weeks before surgery
  Interventions: Drug: Cholecalciferol
- Vitamin D deficiency observation (No Intervention): subjects with 25OHD < 20 ng/mL that will not receive cholecalciferol before surgery
- Vitamin D sufficiency (No Intervention): controls with 25OHD >= 20 ng/mL that will not receive cholecalciferol before surgery

INTERVENTIONS:
Drug: Cholecalciferol — 100,000 U of cholecalciferol weekly for 4 weeks
  Arms: Vitamin D deficiency treatment

SUMMARY:
Hypocalcemia is a frequent adverse event after thyroidectomy. It is usually related to hypoparathyroidism, but preoperative hypocalcemia, hypomagnesemia or vitamin D deficiency contributes to it. This study aims to determine the frequency of vitamin D deficiency or insufficiency in patients submitted to thyroidectomy, to define the risk attributed to vitamin D deficiency to postoperative hypocalcemia, to identify other factors associated to postoperative calcium disorder, and to evaluate the benefit of preoperative treatment of vitamin D deficiency to prevent postoperative hypocalcemia.

DETAILED DESCRIPTION:
Subjects to be submitted to total thyroidectomy will be included in the study. The investigators will evaluate serum levels of total calcium, ionic calcium, phosphorus, magnesium, creatinine, albumin, alkaline phosphatase, fasting glucose, thyroid stimulating hormone (TSH), free thyroxin (FT4), intact parathyroid hormone (PTH), 25 hydroxy vitamin D (25OHD), osteocalcin, C-terminal telopeptide (CTX) and procollagen type 1 amino-terminal propeptide (P1NP). Patients will be randomized to 3 groups: (1) 30 subjects with 25OHD < 20 ng/mL that will receive 100,000U of cholecalciferol weekly for 4 weeks before surgery, (2) 30 subjects with 25OHD < 20 ng/mL that will not receive cholecalciferol before surgery and (3) 30 controls with 25OHD >= 20 ng/mL that will not receive cholecalciferol before surgery. Afterwards, the investigators will evaluate immediate postoperative PTH and measure serum levels of total calcium, ionic calcium, magnesium, alkaline phosphatase, osteocalcin, CTX and P1NP in first and second postoperative days for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients that will be submitted to total thyroidectomy

Exclusion Criteria:

* < 18 year-old
* chronic renal failure (creatinine > 1.5 mg/dL)
* fasting glucose > 200 mg/dl
* albumin < 3.5 g/L
* preoperative use of calcium supplements, bisphosphonates, corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
postoperative hypocalcemia | up to 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Debora LS Danilovic, M.D., PhD., Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil